CLINICAL TRIAL: NCT07293871
Title: Ultrasound Neuroimmune Modulation in Adults With Rheumatoid Arthritis: Feasibility and Safety in a Multicenter, Randomized, Double-Blind, Sham-Controlled Trial
Brief Title: Ultrasound Neuroimmune Modulation in Adults With Rheumatoid Arthritis
Acronym: SUSTAIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Surf Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SURF-CLN-003
Record Dates: First submitted 2025-12-02; First posted 2025-12-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: rheumatoid arthritis; RA; noninvasive; autoimmune
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Stage 1 is a single group and open-label. Stage 2 is randomized, double-blind, sham-controlled with 2 treatment arms, active and sham, that are allocated 2:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In addition the laboratory personnel analyzing the blood samples, and the statistician analyzing the trial data will be blinded to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Daily active stimulation for 8 weeks
  Interventions: Device: Active treatment
- Control (Sham Comparator): Daily sham stimulation, for 8 weeks, which will look and feel the same as active stimulation, but with no ultrasound energy entering the body
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Active treatment — Daily active ultrasound stimulation
  Arms: Treatment
Device: Sham (No Treatment) — Daily sham ultrasound stimulation
  Arms: Control

SUMMARY:
This two-stage, multicenter clinical trial is designed to evaluate the feasibility, safety, and preliminary efficacy of at-home ultrasound stimulation to activate immune-neuromodulation in patients with rheumatoid arthritis (RA) and at least moderate disease activity. The study will enroll up to 40 participants at up to 6 sites across 2 stages. The findings from this trial will directly inform the design and power calculations for a future pivotal trial by identifying an appropriate effect size and confirming protocol feasibility and safety for a daily home-use therapy.

DETAILED DESCRIPTION:
Stage 1 is an open-label pilot study of 5-8 participants receiving active daily ultrasound stimulation for 8 weeks. The primary objective is to assess feasibility and safety, defined by the absence of device-related serious adverse events (SAEs) or Grade ≥2 adverse events (AEs) requiring medical intervention per CTCAE criteria. Data from Stage 1 will be used to refine trial procedures and confirm readiness for Stage 2.

Stage 2 consists of a randomized double-blind, sham-controlled study enrolling up to 30 participants, allocated 2:1 to receive active or sham daily ultrasound stimulation for 8 weeks. This stage is designed to estimate the treatment effect size, using clinical and biomarker-based endpoints, and to collect safety and adherence data on a larger cohort.

All participants will be followed through Week 12 to assess post-treatment safety and durability of clinical and immunologic effects.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosis of rheumatoid arthritis as defined by ACR/EULAR 2010 classification criteria
* A positive test result for Rheumatoid Factor (RF) > 14 IU/mL and/or Anti-Citrullinated Protein Antibodies (Anti-CCP) ≥ 20 U/mL
* At least moderate disease activity, defined as DAS28-CRP > 3.8 and at least 4/28 tender and 4/28 swollen joints at the screening and baseline visits
* High sensitivity CRP (hsCRP) ≥ 10 mg/L at the screening and baseline visits
* On stable dose of background DMARD therapy (see exclusion criteria)
* Able and willing to comply with all study-related procedures, including at-home device use, daily treatment, scheduled visits, and assessments

Exclusion Criteria:

* Unable to provide informed consent
* Current or planned participation in another interventional clinical trial
* Prior use of > 2 biologic or targeted synthetic DMARDs for RA where the primary reason for discontinuation was efficacy
* Conventional synthetic DMARDs:

  * Initiated within last 12 weeks or adjusted dose within 4 weeks prior to enrollment
  * Inability to maintain a stable dose during the study
* Biologic DMARDs:

  * Initiated or dose-adjusted within 12 weeks prior to enrollment
  * Inability to maintain a stable dose during the study
* JAK inhibitors:

  * Use within 4 weeks prior to enrollment or expected use during study participation
* Corticosteroids:

  * Initiated or dose-adjusted within 4 weeks prior to enrollment
  * Current dose > 10 mg/day prednisone (or equivalent)
* Current tobacco or nicotine product use
* Pregnant or planning to become pregnant during the study period
* Known hypersensitivity to ultrasound gel or membrane components
* Active bacterial, viral, or fungal infection
* Receiving chemotherapy or immunotherapy for malignancy
* History of splenic disorders, including splenectomy, congenital asplenia, or splenomegaly on screening ultrasound
* Rash, wound, or skin infection overlying the spleen
* History of vagal nerve injury, vagotomy, or known autonomic neuropathy
* Recent abdominal surgery or trauma within 30 days of screening
* Uncontrolled fibromyalgia or other diffuse pain syndromes that may confound symptom reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in high sensitivity CRP (hsCRP) | 8 weeks
  The primary endpoint is the change in hsCRP from baseline to weeks 2, 4, 6 and 8. The baseline value will be calculated as the average of the screening and baseline visits, both of which must be ≥ 10 mg/L.
Incidence of Adverse Events | 12 weeks
  All adverse events (AEs) regardless of treatment group that occur over the 12 week enrollment period will be coded and summarized by frequency, severity, and relatedness using the latest MedDRA version (v28.1).

SECONDARY OUTCOMES:
American College of Rheumatology (ACR) 20, 50 and 70 response rates | Week 8
  Difference between treatment and control groups in the proportion of subjects who achieve at least 20%, 50%, and 70% improvement from baseline to Week 8 in tender and swollen joint counts of 28 joints (scale 0=best to 28=worst) and 3 out of the following 5 measures: Health Assessment Questionnaire Disability Index (HAQ-DI) score (scale 0=no difficulty to 3=unable to do), subject global assessment (0=best to 10=worst), subject pain (0=no pain to 10=worst), evaluator's global assessment (0=best to 10=worst), or high sensitivity C-reactive protein (hsCRP) concentration (mg/mL).
Change in Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP). | Week 8
  Defined by EULAR based on a composite score of 4 items: tender and swollen joint counts of 28 joints (scale 0=best to 28=worst), subject global assessment (0=best to 10=worst) and high-sensitivity C-reactive protein (hsCRP) concentration (mg/L). DAS28-CRP response based on the minimal clinically important difference (MCID) of -1.2 from baseline to week 8.
Change in Heath Assessment Questionnaire Disability Index (HAQ-DI) | Week 8
  Haq-DI assesses physical function through eight daily activity domains (scale 0=no difficulty to 3=unable to do). Change from baseline to week 8 based on the MCID of -0.22.
Change in Clinical Disease Activity Index (CDAI) score for Rheumatoid Arthritis | Week 8
  The CDAI assesses disease activity by summing tender joint count (TJC), swollen joint count (SJC), patient global assessment (PGA), and physician global assessment (EGA). CDAI will be assessed from Baseline to Week 8.
Change in Simplified Disease Activity Index (SDAI) for Rheumatoid Arthritis (RA) | Week 8
  The SDAI is a measure of disease activity that includes all the 4 components of the CDAI, plus CRP. SDAI will be assessed from baseline to Week 8.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Precision Comprehensive Clinical Research Solutions, Irving, Texas

IPD SHARING:
Plan to Share IPD: No